CLINICAL TRIAL: NCT05077787
Title: Tactile and Kinaesthetic Stimulation in Preterm Neonates With Hyperbilirubinaemia
Brief Title: Tactile and Kinaesthetic Stimulation in Neonates With Hyperbilirubinaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1269-9921
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Neonates recruited in experimental group will receive massage therapy and kinaesthetic stimulation for 15 minutes along with phototherapy for consecutive days . It will be given in three phases first massage therapy will be given for 5 minutes, followed by movement of limbs for 5 minutes and then again massage therapy will be repeated for 5 minutes.
  Interventions: Other: Massage therapy; Other: Kinaesthetic stimulation
- Control Group (No Intervention): Neonates recruited in control group will receive phototherapy alone along with regular care

INTERVENTIONS:
Other: Massage therapy — Massage therapy includes stroking, kneading, rolling, tapping, vibration and effleurage over the face, chest ,abdomen and back. Massage therapy will be given for 5 minutes and will be repeated twice.
  Arms: Experimental Group
Other: Kinaesthetic stimulation — Kinaesthetic stimulation includes passive flexion and extension movements of shoulder joint, elbow joint, hip joint, knee joint and both lower limbs together. It will be given for 5 minutes in each intervention
  Arms: Experimental Group

SUMMARY:
Hyperbilirubinemia is the most common problem seen in neonates, owing to severe complications in their lifetime. The study design of the study is pretest - a posttest experimental design. Criterion-based purposive sampling will be used for recruiting the neonates. In the study neonates will be selected according to the selection criteria and will be allocated into two groups using computer-based randomization.The Intervention group - neonates will receive tactile and kinesthetic stimulation for 15 minutes for 3 consecutive days, 1 hour after feeding twice daily along with Phototherapy, Control group - Phototherapy alone will be given along with conventional NICU care. Total serum bilirubin will be assessed as outcome measures daily once. Transcutaneous bilirubin will be assessed after every intervention.

ELIGIBILITY:
1. New born in Neonatal Intensive Care Unit
2. Stable vitals
3. Full Term and Preterm neonates
4. Gestational age 34 weeks to 40 weeks
5. Birth weight -1800 - 3000 g
6. APGAR Score at birth of 8 -10
7. Total serum bilirubin levels > 10 mg/dL

Ages: 24 Hours to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Total Serum Bilirubin (TSB) | Changes in the Total Serum Bilirubin level will be measured at baseline and at the end of three days intervention
  It will measure total bilirubin level in blood of neonates
Transcutaneous Bilirubin (TcB) | Changes in the Transcutaneous Bilirubin level will be measured daily for three days before and after intervention
  Transcutaneous Bilirubin will measure neonatal jaundice.
Weight Gain | Changes in the weight will be measured at baseline and at the end of three days intervention
  Weight gain will evaluate the change in neonatal weight

CONTACTS AND LOCATIONS:
Overall Officials: Saumya Kothiyal, MPT, Principal Investigator — Maharishi Markendeshawar (Deemed to be University)
Locations (1):
- Civil Hospital, Ropar, Punjab, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahmawati D, Sampurna MTA, Etika R, Utomo MT, Bos AF. Transcutaneous bilirubin level to predict hyperbilirubinemia in preterm neonates. F1000Res. 2020 Apr 28;9:300. doi: 10.12688/f1000research.22264.2. eCollection 2020. PMID 33014346
- [Background] Lin CH, Yang HC, Cheng CS, Yen CE. Effects of infant massage on jaundiced neonates undergoing phototherapy. Ital J Pediatr. 2015 Nov 25;41:94. doi: 10.1186/s13052-015-0202-y. PMID 26607061
- [Background] Field T. Pediatric Massage Therapy Research: A Narrative Review. Children (Basel). 2019 Jun 6;6(6):78. doi: 10.3390/children6060078. PMID 31174382
- [Background] Niemi AK. Review of Randomized Controlled Trials of Massage in Preterm Infants. Children (Basel). 2017 Apr 3;4(4):21. doi: 10.3390/children4040021. PMID 28368368